CLINICAL TRIAL: NCT06345248
Title: Laparoscopic-assisted Versus Ultrasonography-guided Transversus Abdominis Plane Block in Laparoscopic Sleeve Gastrectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-854
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Transversus Abdominis Plane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-TAP group (Active Comparator)
  Interventions: Procedure: US-TAP
- LAPTAP group (Active Comparator)
  Interventions: Procedure: LAPTAP

INTERVENTIONS:
Procedure: US-TAP — regional block team under ultrasound guidance
  Arms: US-TAP group
Procedure: LAPTAP — performed TAP block under direct visualization with the laparoscope
  Arms: LAPTAP group

SUMMARY:
The transversus abdominis plane (TAP) block, whereby local anesthetic is injected between the internal oblique and transversus abdominis fascia to facilitate blockade of somatic afferents nerves, is an effective, non-narcotic adjunct incorporated into many ERAS protocols. We hypothesized that surgeon delivered LAP-TAPs would be non-inferior to anesthesia-delivered US-TAPs in terms of post-operative pain control

ELIGIBILITY:
Inclusion Criteria:

Elective laparoscopic sleeve gastrectomy aging > 18years BMI > 40 kg/m2, ASA score I-III

Exclusion Criteria:

history of chronic opioid consumption suffering from contraindications to regional blocks suffering from allergy to study drugs, history of prior complex abdominal wall reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
morphine needed | UP TO 24 HOURE
  mg

SECONDARY OUTCOMES:
first analgesic request time | up to 24 hours
  he time elapsed between the end of the operation till the first analgesic dose
patients' satisfaction | UP TO 24 HOURE
  scale of 1-4 (1, poor; 2, acceptable; 3, satisfactory; and 4, excellent)
opioid-associated side effects | UP TO 24 HOURE
  bradycardia and hypotesion

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Still working